CLINICAL TRIAL: NCT01223274
Title: Delivery Room Continuous Positive Airway Pressure/Positive End Expiratory Pressure (CPAP/PEEP) in Extremely Low Birth Weight (ELBW) Infants
Brief Title: Delivery Room CPAP in Extremely Low Birth Weight Infants
Acronym: DR-CPAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Neil N. Finer, Lead Principal Investigator, University of California - San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0028; U10HD021364 (NIH); M01RR000080 (NIH); U10HD034216 (NIH); U10HD027853 (NIH); M01RR008084 (NIH); U10HD021397 (NIH); M01RR016587 (NIH); U10HD040461 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Bronchopulmonary Dysplasia; Continuous Positive Airway Pressure
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Very Low Birth Weight (VLBW); Prematurity; Mechanical ventilation; Positive-Pressure Ventilation; Surfactant; Intubation; Pulse oximetry; Oxygen saturation
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP/PEEP Intervention (Experimental): Infants received 100% oxygen by facemask and continuous positive airway pressure (CPAP) or positive pressure ventilation (PPV) with positive end-expiratory pressure (PEEP), if the infant required PPV.
  Interventions: Device: CPAP/PEEP
- Control (Active Comparator): Control infants were treated with 100% oxygen and no CPAP. When a control infant required PPV, no PEEP was used.
  Interventions: Device: Standard management practices

INTERVENTIONS:
Device: CPAP/PEEP — Infants received 100% oxygen by facemask and continuous positive airway pressure (CPAP) or positive pressure ventilation (PPV) with positive end-expiratory pressure (PEEP), if the infant required PPV.
  Other Names: Neopuff
  Arms: CPAP/PEEP Intervention
Device: Standard management practices — Control infants were treated with 100% oxygen and no CPAP. When a control infant required PPV, no PEEP was used.
  Arms: Control

SUMMARY:
This pilot study was designed to determine the feasibility of randomizing extremely low birth weight (ELBW) infants <28 weeks' gestation who required resuscitation to one of two resuscitation methods, either: (a) 100% oxygen by facemask and continuous positive airway pressure (CPAP) or positive pressure ventilation (PPV) with positive end-expiratory pressure (PEEP), if the infant required PPV (the intervention group); or (b) 100% oxygen and no CPAP and no PEEP if the infant required PPV (the control group).

DETAILED DESCRIPTION:
Previous studies suggested that early continuous airway positive pressure (CPAP) may be beneficial in reducing ventilator dependence and subsequent bronchopulmonary dysplasia (BPD) in extremely low birth weight (ELBW) infants. These studies did not test for the optimal timing of CPAP initiation or compare CPAP/PEEP initiation in the delivery room against standard resuscitation methods. Current practice at the time was for the ELBW infant to be intubated early and administered prophylactic surfactant. The feasibility of initiating CPAP in the DR and continuing this therapy without intubation for surfactant had not been determined prospectively in a population of ELBW infants.

This pilot study was designed to determine the feasibility of randomizing extremely low birth weight (ELBW) infants <28 weeks' gestation who required resuscitation to one of two resuscitation methods, either: (a) 100% oxygen by facemask and continuous positive airway pressure (CPAP) or positive pressure ventilation (PPV) with positive end-expiratory pressure (PEEP), if the infant required PPV (the intervention group); or (b) 100% oxygen and no CPAP and no PEEP if the infant required PPV (the control group).

ELIGIBILITY:
Inclusion Criteria:

* Infants delivered in a specially equipped resuscitation room(s)
* <28 weeks gestational age by best obstetric estimate before delivery
* Requiring resuscitation

Exclusion Criteria:

* No known major congenital anomalies
* Decision made not to provide full resuscitation

Max Age: 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2002-07; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Compliance with the study protocol | 6 months

SECONDARY OUTCOMES:
Extent of resuscitation needed | Until admission to NICU
Five minute Apgar | 5 minutes after birth
Total duration of mechanical ventilation | Until hospital discharge or 120 days of life
Proportion of infants requiring surfactant | 1 day of life
Bronchopulmonary dysplasia (BPD) | 36 weeks of life
Number and duration of intubation attempts | Until admission to the NICU
Infants who required positive pressure ventilation for resuscitation in the DR/resuscitation room | Until admission to the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Neil N. Finer, MD, Study Director — University of California, San Diego; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies & Children's Hospital; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Charles R. Bauer, MD, Principal Investigator — University of Miami; W. Kenneth Poole, PhD, Principal Investigator — RTI International
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Diego, San Diego, California
  - University of Miami, Miami, Florida
  - RTI International, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio

REFERENCES:
- [Result] Finer NN, Carlo WA, Duara S, Fanaroff AA, Donovan EF, Wright LL, Kandefer S, Poole WK; National Institute of Child Health and Human Development Neonatal Research Network. Delivery room continuous positive airway pressure/positive end-expiratory pressure in extremely low birth weight infants: a feasibility trial. Pediatrics. 2004 Sep;114(3):651-7. doi: 10.1542/peds.2004-0394. PMID 15342835
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/